CLINICAL TRIAL: NCT06349915
Title: A Pilot Evaluation of a Digital Peer Support Intervention for Suicidal Adolescents
Acronym: SWEEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: American Foundation for Suicide Prevention (Other); Yeshiva University (Other); Ilumivu (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023-15217
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Suicide
Keywords: digital intervention; community participation; ecological momentary assessment
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Intervention Model Description: The first 6 participants will serve as a brief pilot to validate outcomes and the acceptability of the intervention. The study team may make slight changes to the intervention (e.g., time of day the suicide recovery narratives are administered, or which narratives are presented) before recruiting the remaining 40 participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): This is a single-arm study. All participants will be allocated to the intervention arm, in which they will receive the digital narrative therapy.
  Interventions: Behavioral: Supporting Wellbeing with Everyday Experiences of Peers (SWEEP)

INTERVENTIONS:
Behavioral: Supporting Wellbeing with Everyday Experiences of Peers (SWEEP) — Each day during a 14-day trial period, participants will receive one narrative featuring lived experience with and recovery from suicidal thoughts and behaviors. These narratives will be presented in audio and text format via a smartphone app. Participants will also complete self-report surveys assessing study outcomes using the same smartphone app five times per day.
  Other Names: SWEEP

SUMMARY:
Suicide risk has increased among youth in underserved communities, where access to mental healthcare is limited. To address this need, the investigator team plans to evaluate the preliminary efficacy of a brief, low-cost, culturally responsive digital intervention for ethnically diverse youth at risk for suicide in The Bronx, New York. In collaboration with community stakeholders, suicide recovery narratives, featuring adolescents' experiences related to recovery from suicidal thoughts will be developed. A smartphone ecological momentary assessment (EMA) app will be used to evaluate whether a curriculum of these narratives provides anti-suicidal benefits to at-risk adolescents.

DETAILED DESCRIPTION:
This is a single-arm investigation of a novel suicide prevention intervention, called "Supporting Wellbeing with Everyday Experiences of Peers" (SWEEP). In a preliminary phase (Phase 1) of the study, suicide recovery narratives: short first-person stories about lived experience with and recovery from Bronx Adolescents will be collected. The investigator team will then evaluate evaluate the anti-suicidal benefits of this intervention in a single-arm trial. In a subsequent phase (Phase 2), adolescent participants (n=46) will be provided with the SWEEP intervention, which involves reading or listening to one suicide recovery narrative each day during the 14-day trial. Six of the 46 participants will be adolescents, with recent suicidal thoughts or depression, who are currently receiving mental healthcare in Montefiore's Outpatient Psychiatry Department, rather than those on the waitlist to receive these services. All six participants will then complete a post-intervention qualitative interview to inform potential changes to intervention procedures. During this second phase, suicide recovery narratives will be provided, in audio and text formats, via a smartphone app. That same smartphone app will also collect real-time (ecological momentary) assessments of suicidal thoughts, as well as secondary and additional outcomes, five times per day. The investigator team will evaluate whether participants experience reductions in the intensity of suicidal thoughts over the course of the 14-day trial. During Phase 3, participants will be recruited to a control condition (n=15) and a treatment condition (n=30). Those in the Phase 3 treatment condition will receive the same intervention (1 SWEEP narrative per day for 14 days + 3x/day EMA) as those in Phase 2. Those in the Control condition will receive 3x/day EMA only.

ELIGIBILITY:
Inclusion Criteria:

* past-month history of suicidal thoughts
* past-month history of Major depressive disorder
* possession of apple or android smartphone with data plan

Exclusion Criteria:

* inability to read/write in English
* Active mania
* Active psychosis
* Autism spectrum disorder

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Suicidal Thoughts | 5 times per day during 14-day trial
  Participants will self-report their current subjective intensity of suicidal thoughts using an 11-point Likert-type scale, with higher scores indicating more intense suicidal thoughts.

SECONDARY OUTCOMES:
Suicidal Urge Resistance | 5 times per day during 14-day trial
  Participants will self-report the strength of their current ability to resist suicidal urges using an 11-point Likert-type scale, with higher scores indicating greater ability to resist suicidal urges.
Social Connectedness | 5 times per day during 14-day trial
  Participants will self-report their current feelings of being connected to other people using an 11-point Likert-type scale, with higher scores indicating feeling more being connected to other people.
Optimism | 5 times per day during 14-day trial
  Participants will self-report their current of feelings of optimism about the future using an 11-point Likert-type scale, with higher scores indicating greater optimism.
Social Support | 5 times per day during 14-day trial
  Participants will self-report their current perception of the availability of emotional support from others using an 11-point Likert-type scale, with higher scores indicating the perception greater availability of emotional support from others.
Intervention Acceptability | Study conclusion (at the end of the 14-day trial)
  Participants will self-report their current perception of acceptability of the SWEEP intervention across three items. Participants will rate the usefulness of receiving the narratives using a 7-point Likert-type scale, with higher scores indicating that the narratives were more useful. Participants will rate the difficulty of reading or listening to the narratives each day using a 7-point Likert-type scale, with higher scores indicating that the narratives were more difficult to read or listen to. This item will be reverse coded. Participants will rate how willing they are to recommend the narratives to their peers using a 7-point Likert-type scale, with higher scores indicating greater willingness to recommend the narratives. Each of these items will be evaluated in isolation, as well as in aggregate using both summation and an arithmetic mean score.

OTHER OUTCOMES:
Emotions | 5 times per day during 14-day trial
  Participants will self-report the current intensity of 10 emotions: excited, guilty, scared, proud, irritated, ashamed, inspired, nervous, determined, angry. Each emotion will be rated on an 11-point Likert-type scale with higher scores indicating more intense emotion. Each of these items will be evaluated in isolation, as well as in aggregate using arithmetic mean. For aggregating an overall emotion score, the positive emotions excited, proud, inspired, and determined will be reverse-scored to provide an aggregate rating of negative emotion.
Treatment Readiness | Baseline (prior to starting the 14-day trail) and study conclusion (at the end of the 14-day trial)
  Participants will self-report their current readiness for mental health treatment across 4 items. Participants will rate their motivation for beginning regular mental health services using a 7-point Likert-type scale, with higher scores indicating greater readiness to begin regular services. Participants will rate their anxiety about discussing personal difficulties with a mental health professional using a 7-point Likert-type scale, with higher scores indicating greater anxiety. This item will be reverse coded. Participants will rate how confident they feel that regular mental health services will be helpful using a 7-point Likert-type scale, with higher scores indicating greater confidence. Participants will rate how necessary they feel that regular mental health services are for them using a 7-point Likert-type scale, with higher scores indicating greater feelings of necessity. Each item will be evaluated in isolation and in aggregate using both summation and arithmetic mean score.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Franz, Ph.D., Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Health System, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
The research team will consider requests to share specific data with qualified research teams upon request

REFERENCES:
- [Background] Franz PJ, Mou D, Kessler DT, Stubbing J, Jaroszewski AC, Ray S, Cao-Silveira VB, Bachman S, Schuster S, Graupensperger D, Alpert JE, Porath M, Nock MK. Digital bibliotherapy as a scalable intervention for suicidal thoughts: A randomized controlled trial. J Consult Clin Psychol. 2022 Aug;90(8):626-637. doi: 10.1037/ccp0000752. PMID 36066864
- [Background] Centers for Disease Control and Prevention. 10 leading causes of death, United States. WISQARS Fatal Injury Data Visualization Tool.
- [Background] Fox KR, Huang X, Guzman EM, Funsch KM, Cha CB, Ribeiro JD, Franklin JC. Interventions for suicide and self-injury: A meta-analysis of randomized controlled trials across nearly 50 years of research. Psychol Bull. 2020 Dec;146(12):1117-1145. doi: 10.1037/bul0000305. Epub 2020 Oct 29. PMID 33119344
- [Background] Alvarez K, Polanco-Roman L, Samuel Breslow A, Molock S. Structural Racism and Suicide Prevention for Ethnoracially Minoritized Youth: A Conceptual Framework and Illustration Across Systems. Am J Psychiatry. 2022 Jun;179(6):422-433. doi: 10.1176/appi.ajp.21101001. PMID 35599542
- [Background] Bray MJC, Daneshvari NO, Radhakrishnan I, Cubbage J, Eagle M, Southall P, Nestadt PS. Racial Differences in Statewide Suicide Mortality Trends in Maryland During the Coronavirus Disease 2019 (COVID-19) Pandemic. JAMA Psychiatry. 2021 Apr 1;78(4):444-447. doi: 10.1001/jamapsychiatry.2020.3938. PMID 33325985
- [Background] Weimerskirch PJ. Benjamin Rush and John Minson Galt, II. Pioneers of bibliotherapy in America. Bull Med Libr Assoc. 1965 Oct;53(4):510-26. PMID 5319266
- [Background] Stip E, Ostlundh L, Abdel Aziz K. Bibliotherapy: Reading OVID During COVID. Front Psychiatry. 2020 Dec 7;11:567539. doi: 10.3389/fpsyt.2020.567539. eCollection 2020. PMID 33364987
- [Background] Evans K, Tyrer P, Catalan J, Schmidt U, Davidson K, Dent J, Tata P, Thornton S, Barber J, Thompson S. Manual-assisted cognitive-behaviour therapy (MACT): a randomized controlled trial of a brief intervention with bibliotherapy in the treatment of recurrent deliberate self-harm. Psychol Med. 1999 Jan;29(1):19-25. doi: 10.1017/s003329179800765x. PMID 10077290
- [Background] Gualano MR, Bert F, Martorana M, Voglino G, Andriolo V, Thomas R, Gramaglia C, Zeppegno P, Siliquini R. The long-term effects of bibliotherapy in depression treatment: Systematic review of randomized clinical trials. Clin Psychol Rev. 2017 Dec;58:49-58. doi: 10.1016/j.cpr.2017.09.006. Epub 2017 Sep 29. PMID 28993103
- [Background] Bietti LM, Tilston O, Bangerter A. Storytelling as Adaptive Collective Sensemaking. Top Cogn Sci. 2019 Oct;11(4):710-732. doi: 10.1111/tops.12358. Epub 2018 Jun 28. PMID 29954043
- [Background] Rennick-Egglestone S, Morgan K, Llewellyn-Beardsley J, Ramsay A, McGranahan R, Gillard S, Hui A, Ng F, Schneider J, Booth S, Pinfold V, Davidson L, Franklin D, Bradstreet S, Arbour S, Slade M. Mental Health Recovery Narratives and Their Impact on Recipients: Systematic Review and Narrative Synthesis. Can J Psychiatry. 2019 Oct;64(10):669-679. doi: 10.1177/0706743719846108. Epub 2019 May 2. PMID 31046432
- [Background] Van Orden KA, Witte TK, Cukrowicz KC, Braithwaite SR, Selby EA, Joiner TE Jr. The interpersonal theory of suicide. Psychol Rev. 2010 Apr;117(2):575-600. doi: 10.1037/a0018697. PMID 20438238
- [Background] Joiner T. Why People Die by Suicide. Harvard University Press; 2005.
- [Background] Nock MK, Green JG, Hwang I, McLaughlin KA, Sampson NA, Zaslavsky AM, Kessler RC. Prevalence, correlates, and treatment of lifetime suicidal behavior among adolescents: results from the National Comorbidity Survey Replication Adolescent Supplement. JAMA Psychiatry. 2013 Mar;70(3):300-10. doi: 10.1001/2013.jamapsychiatry.55. PMID 23303463
- [Background] Millner AJ, Lee MD, Nock MK. Describing and Measuring the Pathway to Suicide Attempts: A Preliminary Study. Suicide Life Threat Behav. 2017 Jun;47(3):353-369. doi: 10.1111/sltb.12284. Epub 2016 Aug 1. PMID 27477787
- [Background] Franklin JC, Ribeiro JD, Fox KR, Bentley KH, Kleiman EM, Huang X, Musacchio KM, Jaroszewski AC, Chang BP, Nock MK. Risk factors for suicidal thoughts and behaviors: A meta-analysis of 50 years of research. Psychol Bull. 2017 Feb;143(2):187-232. doi: 10.1037/bul0000084. Epub 2016 Nov 14. PMID 27841450
- [Background] Roswarski T, Dunn J. The Role of Help and Hope in Prevention and Early Intervention with Suicidal Adolescents: Implications for Mental Health Counselors. J Ment Health Couns. 2009;31(1):34-46. doi:10.17744/mehc.31.1.u150745762627518
- [Background] Franz PJ, Nook EC, Mair P, Nock MK. Using Topic Modeling to Detect and Describe Self-Injurious and Related Content on a Large-Scale Digital Platform. Suicide Life Threat Behav. 2020 Feb;50(1):5-18. doi: 10.1111/sltb.12569. Epub 2019 Jul 2. PMID 31264733